CLINICAL TRIAL: NCT03057015
Title: Addition of Clonidine to Ropivacaine in Adductor Canal Block for Postoperative Pain Relief in Total Knee Arthroplasty: A Prospective Randomized Double Blind Placebo Controlled Trial
Brief Title: Addition of Clonidine to Ropivacaine in Adductor Canal Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Borzoo Farhang, Clinical Instructor of Anesthesiology, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHRMS 17-0107
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Clonidine; Ropivacaine; Dexamethasone; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clonidine (Experimental): 50 mcg clonidine + 0.5% ropivacaine + 2 mg dexamethasone + 5 mcg/ml epinephrine in 20 ml solution
  Interventions: Drug: Clonidine; Drug: Ropivacaine; Drug: Dexamethasone; Drug: Epinephrine
- Placebo (Placebo Comparator): 0.5 ml normal saline + 0.5% ropivacaine + 2 mg dexamethasone + 5 mcg/ml epinephrine in 20 ml solution
  Interventions: Drug: Placebo; Drug: Ropivacaine; Drug: Dexamethasone; Drug: Epinephrine

INTERVENTIONS:
Drug: Clonidine — 50 mcg Clonidine added to the solution of 0.5% ropivacaine, 2 mg dexamethasone and 5 mcg/ml epinephrine for adductor canal block-present in the treatment group.
  Arms: Clonidine
Drug: Placebo — Normal saline added to the solution of 0.5% ropivacaine, 2 mg dexamethasone and 5 mcg/ml epinephrine for adductor canal block-present in the placebo group.
  Arms: Placebo
Drug: Ropivacaine — Clonidine or Placebo added to the solution of 0.5% ropivacaine, 2 mg dexamethasone and 5 mcg/ml epinephrine for adductor canal block-present in both treatment and placebo groups.
Drug: Dexamethasone — Clonidine or Placebo added to the solution of 0.5% ropivacaine, 2 mg dexamethasone and 5 mcg/ml epinephrine for adductor canal block-present in both treatment and placebo groups.
Drug: Epinephrine — Clonidine or Placebo added to the solution of 0.5% ropivacaine, 2 mg dexamethasone and 5 mcg/ml epinephrine for adductor canal block-present in both treatment and placebo groups.

SUMMARY:
Total knee arthroplasty (knee replacement) is a common orthopedic procedure for osteoarthritis. This procedure is performed either under general anesthesia or spinal anesthesia; after the procedure in the recovery room, these patients undergo adductor canal block, which is a nerve block to provide 8-14 hours of postoperative pain control. For this nerve block, 15-20 ml of local anesthetic is combined with adjuvant medications to improve the quality of pain control as well as the duration of pain relief. The primary local anesthetic used for adductor canal block is ropivacaine, and the commonly used adjuvants are epinephrine and dexamethasone.

There is conflicting data available in the literature regarding efficacy of addition of clonidine to the local anesthetic injection in peripheral nerve blocks, and there is no data assessing the efficacy of this medication in adductor canal blocks.

Once the consent process is completed, patients are enrolled in two arms. Upon conclusion of surgery, a sealed and coded envelope with either clonidine or the placebo syringe will be given to the acute pain service staff performing the nerve block. This will be mixed with local anesthetic solution and injected in the adductor canal under ultrasound guidance.

The primary outcome measure will be the duration of analgesia, which will be assessed as the time interval between placement of adductor canal block to the first request of opioid analgesic by patients (which will be obtained from hospital electronic medical records). Secondary outcomes will include:

1. Duration of sensory block, which will be assessed as the time interval between injection of local anesthetic and report of postoperative pain of 3 or more on an 11 point scale (0=no pain; 10= worst pain imaginable) by the patient (this will be assessed every 4 hours).
2. Duration of motor block, which will be assessed as the time interval between the onset of motor block to complete recovery of motor block by assessing straight leg raise strength (this will be assessed every 4 hours).
3. Cumulative 24 and 48 hour opioid analgesic use.
4. Post-block pain scores, evaluated by an 11 point pain score (0-10), which will be done every 15 minutes for the first hour after surgery and every 4 hours thereafter for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 and older
* ASA physical status classification system I, II and III (healthy patient or patient with mild to moderate systemic disease)
* Patient coming in for elective total knee arthroplasty under general or neuraxial anesthesia and postoperative adductor canal block
* Patients staying for at least 24 hrs post operatively
* Patients who provide informed consent
* Patients presenting for surgery >1 hour in length and <6 hours.

Exclusion Criteria:

* History of recent common colds, upper respiratory infections or immune deficiencies
* Patients allergic to clonidine
* Pregnant women (all women of childbearing age undergo pregnancy testing prior to anesthesia as per UVMMC peri-operative protocol)
* Patients who are already on chronic clonidine therapy for management of blood pressure
* Patients on chronic opioid therapy defined as more than 10 mg of oxycodone per day (or equivalent doses of other opioid analgesics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Duration of Analgesia | 24 hours for primary outcome
  the time interval between placement of adductor canal block to the first request of opioid analgesic by patients

CONTACTS AND LOCATIONS:
Overall Officials: Borzoo Farhang, DO, Principal Investigator — University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided